CLINICAL TRIAL: NCT04986774
Title: Rescue Intracranial Stenting in Acute Ischemic Stroke
Acronym: RISIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Can Tho Stroke International Services Hospital (Other)
Responsible Party: Principal Investigator, Dr. Cuong Tran Chi, Director - Doctor, Can Tho Stroke International Services Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Can Tho SIS Hospital
Record Dates: First submitted 2021-07-11; First posted 2021-08-03 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Acute Stroke; Ischemic Stroke; Intracranial Atherosclerosis; Stent Stenosis; Cerebral Ischemia; Stent Occlusion; Stroke, Ischemic; Intracranial Hemorrhages; Thrombotic Stroke, Acute
Keywords: Acute ischemic stroke; Rescue intracranial stenting; Symptomatic intracerebral hemorrhage; MRI 3 Tesla; Rehabilitation
MeSH Terms: conditions — Stroke; Ischemic Stroke; Intracranial Arteriosclerosis; Brain Ischemia; Intracranial Hemorrhages; Thrombotic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rescue Intracranial Stenting (RIS) (Experimental): RIS in Acute Ischemic Stroke caused by intracranial large vessel occlusion
  Interventions: Procedure: Rescue intracranial stenting

INTERVENTIONS:
Procedure: Rescue intracranial stenting — Rescue Intracranial Stenting in Acute Ischemic Stroke caused by intracranial large vessel occlusion
  Other Names: RIS

SUMMARY:
In acute ischemic stroke caused by intracranial large vessel occlusion, rescue intracranial stenting has been recently a treatment option to achieve recanalization in patients with the failure of mechanical thrombectomy. Nevertheless, there are few studies supporting this beneficial treatment in two cerebral circulations. We aimed to analyse whether the use of rescue intracranial stenting would improve prognosis of patients at 3 months.

DETAILED DESCRIPTION:
In Asia population, large intracranial arterial stenosis lesion accounts for more than 30% in common causes of ischemic stroke, compares with about 10% in Caucasian population every year. Normally, in human brain, there are about 130 billion neurons but they are lost equivalent to their losses in approximately 3.6 years of normal aging in case of a large vessel ischemic stroke untreated each hour. Consequently, after the success of 5 randomized controlled trials about the mechanical thrombectomy, which have been done from December 2010 to December 2014, all of guidelines recommended this technique as the first-line treatment in acute ischemic stroke. However, the HERMES meta-analysis showed that revascularisation failure ratio 28.9% in patients older than 80 years. Recently, in case of mechanical thrombectomy failure, many studies suggested the rescue intracranial stenting could be alternative urgently needed treatment to achieve permanent recanalization which is one of the most important factors impacting on clinical outcomes after acute ischemic stroke. Hence, the aims of our study were to assess both the "non-poor" outcome at 3 months and the symptomatic intracerebral hemorrhage relating to procedure in patients receiving rescue intracranial stenting.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of intracranial large vessel occlusion.
* Absence of intracranial hemorrhage.
* Severe stenosis or reocclusion after mechanical thrombectomy.

Exclusion Criteria:

* Tandem lesion.
* Loss to follow-up after discharge.
* A severe or fatal combined illness before acute ischemic stroke.

Ages: 20 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-05-29 (Actual); Study Completion 2021-08-29 (Actual)

PRIMARY OUTCOMES:
The "non-poor" 3-month outcome rate. | 3 months
  The "non-poor" 3-month outcome rate was accessed by modified Rankin Score (mRS), which comprised of included good (mRS 0 - ≤ 2) and fair (mRS 3).

SECONDARY OUTCOMES:
The symptomatic intracerebral hemorrhage rate. | 24 hours after rescue intracranial stenting.
  The symptomatic intracerebral hemorrhage was defined as patient's intracerebral hemorrhage with postprocedural mRS ≥ 5 and there were no other evident causes for the increased mRS.

CONTACTS AND LOCATIONS:
Overall Officials: Cuong Tran Chi, Doctor, Study Chair — Can Tho SIS Hospital
Locations (1):
- Can Tho SIS Hospital, Can Tho, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stracke CP, Fiehler J, Meyer L, Thomalla G, Krause LU, Lowens S, Rothaupt J, Kim BM, Heo JH, Yeo LLL, Andersson T, Kabbasch C, Dorn F, Chapot R, Hanning U. Emergency Intracranial Stenting in Acute Stroke: Predictors for Poor Outcome and for Complications. J Am Heart Assoc. 2020 Mar 3;9(5):e012795. doi: 10.1161/JAHA.119.012795. Epub 2020 Mar 3. PMID 32122218
- [Background] Perez-Garcia C, Gomez-Escalonilla C, Rosati S, Lopez-Ibor L, Egido JA, Simal P, Moreu M. Use of intracranial stent as rescue therapy after mechanical thrombectomy failure-9-year experience in a comprehensive stroke centre. Neuroradiology. 2020 Nov;62(11):1475-1483. doi: 10.1007/s00234-020-02487-9. Epub 2020 Jun 30. PMID 32607747
- [Background] Alexander MJ, Zauner A, Chaloupka JC, Baxter B, Callison RC, Gupta R, Song SS, Yu W; WEAVE Trial Sites and Interventionalists. WEAVE Trial: Final Results in 152 On-Label Patients. Stroke. 2019 Apr;50(4):889-894. doi: 10.1161/STROKEAHA.118.023996. PMID 31125298
- [Background] Meyer L, Fiehler J, Thomalla G, Krause LU, Lowens S, Rothaupt J, Kim BM, Heo JH, Yeo L, Andersson T, Kabbasch C, Dorn F, Chapot R, Stracke CP, Hanning U. Intracranial Stenting After Failed Thrombectomy in Patients With Moderately Severe Stroke: A Multicenter Cohort Study. Front Neurol. 2020 Feb 14;11:97. doi: 10.3389/fneur.2020.00097. eCollection 2020. PMID 32117041